CLINICAL TRIAL: NCT00917020
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Pilot Study to Evaluate the Efficacy and Safety of Nasal Carbon Dioxide Used As-Needed in the Symptomatic Treatment of Seasonal Allergic Rhinitis
Brief Title: The Effect of Nasal Carbon Dioxide (CO2) Used As-Needed in the Symptomatic Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capnia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C216
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Randomized; Double-Blind; Multi-Center; Phase II; Nasal Carbon Dioxide; Carbon Dioxide; Efficacy; Safety; Total Nasal Symptom Score
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active: CO2 Gas (Experimental)
  Interventions: Drug: Nasal CO2
- Inactive Placebo Gas (Placebo Comparator)
  Interventions: Drug: Inactive Placebo Gas

INTERVENTIONS:
Drug: Nasal CO2 — As-Needed during the 14 day Treatment Period
  Arms: Active: CO2 Gas
Drug: Inactive Placebo Gas — Placebo
  Arms: Inactive Placebo Gas

SUMMARY:
The purpose of this study is to evaluate the effect of as-needed treatment with nasal carbon dioxide in patients with Seasonal Allergic Rhinitis symptoms.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, multi-center, parallel group, pilot study will evaluate the efficacy and safety of as-needed with nasal, non-inhaled administration of CO2 (nasal CO2) in patients with SAR. Approximately 50 patients who meet the eligibility criteria will be enrolled into this study at up to 4 sites to ensure that approximately 30 patients complete the study.

Patients will be randomized to one of two treatment groups and be provided with either an active or placebo dispenser.

All patients will administer study drug for 10 seconds to each nostril once on Day 0 in the clinic then as-needed up to 6 times a day during waking hours (doses must be at least 2 hours apart) for 14 days. Patients will assess their nasal and non-nasal symptoms in a patient diary. Each patient's participation in the study may last up to 72 days.

There will be a total of 5 scheduled clinic visits:

* Visit 1 Screening
* Visit 2 Enrollment (within 42 days of Visit 1)
* Visit 3 Randomization (after the completion of a 3-7 day run-in period)
* Visit 4 Mid-Treatment (Day 7 ± 1 day)
* Visit 5 End of Treatment (within 1-3 days of last study drug administration)

Sites will follow-up with randomized patients via telephone 7 ± 1 days after the last study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be considered eligible for study enrollment:

  * Able to read and understand informed consent form and voluntarily consent to participate in this study by signing the IRB/EC-approved informed consent form
  * Males or females ages 18 - 65 years
  * Able to comply with the requirements of the protocol
  * Minimal 2-year history of seasonal allergic rhinitis requiring pharmacotherapy
  * Positive skin test to one or more seasonal allergens prevalent in the respective local geographical area by either prick or intradermal methods within 12 months prior to enrollment
  * Females of childbearing potential must commit to using an acceptable method of birth control (e.g., oral birth control pills, intrauterine device (IUD), or a double-barrier method of contraception) through 7 days after last study drug administration. To be considered not of childbearing potential, females must be post-menopausal for at least 2 years or be surgically sterile

Exclusion Criteria:

* Patients must not meet any of the following exclusion criteria to be considered eligible for study enrollment:

  * History of asthma (other than mild intermittent)
  * Nasal disorders that are assessed as clinically significant
  * Acute or significant sinusitis or upper respiratory infection within 14 days of enrollment
  * Existing serious medical condition that precludes participation
  * Females who are pregnant or breast-feeding and/or plan to become pregnant or to breast-feed during study participating or within 7 days after last study drug administration
  * Initiation of immunotherapy or have a change in immunotherapy dose within the 6 months preceding enrollment (if on immunotherapy, the same dose must be maintained throughout the trial)
  * Use of medications and/or treatments (e.g., tricyclic antidepressants) that could affect the assessment of the effectiveness of the study drug
  * Use of concomitant medications or other treatments for trigeminally-mediated diseases (i.e., migraine, TMD, trigeminal neuralgia, etc.) for the duration of the Treatment Period of this study
  * An employee of the study site's research department
  * Have a member of the same household also participating in this study
  * Use of any investigational or experimental therapy within 30 days of enrollment
  * Planned travel outside the study area for the duration of study period
  * Participation in a previous study with nasal CO2

Prior to enrollment and the initiation of the run-in period, patients must meet the following criteria:

* Continue to meet all inclusion criteria
* Do not meet any of the exclusion criteria
* Complete the required washout period of the following medications:

  * Nasal or systemic decongestants (3 days)
  * Nasal, ophthalmic, or systemic short-acting antihistamines (7 days)
  * Nasal or systemic long-acting antihistamines such as cetirizine and fexofenadine (7 days)
  * Leukotriene modifiers such as montelukast, zafirlukast and ziluton (7 days)
  * Any other nasal medications including homeopathy, natural products, etc. (7 days)
  * Loratadine (10 days)
  * Nasal cromolyn (14 days)
  * Nasal, inhaled, ophthalmic, or systemic corticosteroids (30 days)
  * Tricyclic antidepressants or any other medication that could affect assessment of the effectiveness of study drug (7 days)

Prior to randomization, patients must meet the following criteria:

* Continue to meet all inclusion criteria
* Do not meet any of the exclusion criteria
* Did not take any medications requiring washout and must agree to refrain from taking any pharmacotherapy or any other treatments for seasonal allergic rhinitis such as homeopathy, natural health products, etc., for their SAR symptoms during the 14-day Treatment Period.
* Complete at least a minimum of symptom score diary entries at the specified timepoints during the baseline symptom assessment period
* Have a minimum total nasal symptom score (TNSS) as defined by the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of as-needed treatment with nasal carbon dioxide (CO2) in patients with seasonal allergic rhinitis (SAR). | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Anish Bhatnagar, MD, Study Director — Capnia, Inc.
Locations (1):
- Capnia Investigative Site, St Louis, Missouri, United States